CLINICAL TRIAL: NCT05013476
Title: Tele-Ultrasound: VIrtual Hands-on Education for Novice Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-3964
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Ultrasound; Education; Virtual
Keywords: tele-education; ultrasound; FAST; Carpal Tunnel
MeSH Terms: conditions — Median Neuropathy

STUDY DESIGN:
Intervention Model Description: Participants will be divided into 2 groups which will experience different experimental conditions.
Masking Description: Participants and staff will be aware of each of the study conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-Person ultrasound participants (Active Comparator): In-Person ultrasound participant's will receive ultrasound training that is guided by online modules (identical to virtual) with trained faculty in the same room with a ration of 4 students to 1 instructor.
  Interventions: Combination Product: Butterfly handheld ultrasound machine
- Virtual ultrasound participants (Active Comparator): Virtual ultrasound participants will receive ultrasound training that is guided by online modules (identical to in-person) with trained faculty present in a private zoom classroom. Faculty will be rotating between breakout rooms and will share the same ratio of participants to staff.
  Interventions: Combination Product: Butterfly handheld ultrasound machine

INTERVENTIONS:
Combination Product: Butterfly handheld ultrasound machine — Both arms of study will utilize the Butterfly ultrasound machine. Only the virtual learners will utilize zoom for their virtual education
  Other Names: Zoom

SUMMARY:
This study is intended to perform a comparative analysis of novice ultrasound users when taught in person versus virtually. This study aims to show that students will not demonstrate a statistical difference in scores learning in in a virtual environment, guided by professionals, when compared to students learning ultrasound in a traditional, in-person format. Utilizing a Butterfly ultrasound machine, a hand held personal ultrasound device, students wil be guided through a FAST (Focused assessment with sonography in trauma) examination and imaging of the carpal tunnel using modules and instructor aid. The FAST (Focused assessment with sonography in trauma) exam images the heart and abdomen for free flowing blood. The carpal tunnel is a region in the wrist that houses the tendons for finger movement. Participants will be assessed on the ability to identify key regions, anatomical landmarks and confidence in utilize the ultrasound machine.

DETAILED DESCRIPTION:
This project intends to adapt previous research ("Innovations with tele-ultrasound in education sonography: the use of tele-ultrasound to train novice scanners") to assess the effectiveness of tele-education using the Butterfly handheld ultrasound device when compared to in person education imaging devices, learning modules and assessments will be kept constant across experimental groups. This experiment aims to adapt the current ultrasound modules used by the University of Colorado Anschutz school of Medicine and Modern Human Anatomy program to formulate in depth modules that outline the following: Carpal Tunnel (wrist), Brachial Plexus (shoulder), and FAST "Focused Assessment with Sonography in Trauma". Additionally, participants will be provided an orientation module that will be completed prior to the live session. Participants will be divided into either the in-person group or virtual group and participate in a live session where participants go through each module with a trained instructor. Participants will be asked to complete a pre/post assessment to determine prior knowledge and the level of learning that took place during the session as well as participant satisfaction and confidence levels.

ELIGIBILITY:
Inclusion Criteria:

* First year medical students enrolled at the University of Colorado, Anschutz Medical Campus with minimal previous ultrasound experience.
* First year graduate students enrolled in the Modern Human Anatomy program (MHA) at the University of Colorado, Anschutz Medical Campus with minimal previous ultrasound experience.

Exclusion Criteria:

* individuals younger than the age of 18.
* individuals not enrolled in the medical school or Modern Human Anatomy program (MHA) programs at Anschutz Medical Campus
* Individuals with greater than minimal ultrasound experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Comparison of participant assesment scores when asked to identify key features of the FAST and Carpal Tunnel between in person learners and virtual learners. | 10 minutes
  Scores are measured on a pass (1) or fail (0) grading system with a total number of 17 points per participant. An Anderson-Darling test will determine if the data is normally distributed. If the data demonstrates normal distribution, either a parametric analysis via a two-way ANOVA or non-parametric equivalent analysis via pairwise Mann-Whitney U will be performed to compare responses from the different groups. Further a Bran-Altman Test will be considered.

SECONDARY OUTCOMES:
Student comparative confidence levels in ultrasound between virtual learners and in-person learners. | 1.5 hours
  Likert Scale measures participant's subjective opinion on a question. Five answer choices are provided on a scale of 0 to 5 with an extreme on both ends, a neutral choice and a middle ground answer for both ends of the spectrum. A higher score represents a greater degree of confidence in the material. Lower scores indicate little to no confidence in the material.
Student comparative satisfaction levels in ultrasound between virtual learners and in-person learners. | 1.5 hours
  Likert Scale measures participant's subjective opinion on a question. Five answer choices are provided on a scale of 0 to 5 with an extreme on both ends, a neutral choice and a middle ground answer for both ends of the spectrum. Higher scores indicate high satisfaction levels with the learning modality. Low scores indicate that participant's did not enjoy the learning modality.

CONTACTS AND LOCATIONS:
Overall Officials: logan T scott, B.S., Principal Investigator — Graduate Student, Masters in Modern Human Anatomy
Locations (1):
- logan T scott, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared with other researchers. Statistical analysis and results will be shared.

REFERENCES:
- [Background] Drake AE, Hy J, MacDougall GA, Holmes B, Icken L, Schrock JW, Jones RA. Innovations with tele-ultrasound in education sonography: the use of tele-ultrasound to train novice scanners. Ultrasound J. 2021 Feb 14;13(1):6. doi: 10.1186/s13089-021-00210-0. PMID 33586112
- [Background] Royer DF, Kessler R, Stowell JR. Evaluation of an innovative hands-on anatomy-centered ultrasound curriculum to supplement graduate gross anatomy education. Anat Sci Educ. 2017 Jul;10(4):348-362. doi: 10.1002/ase.1670. Epub 2016 Nov 21. PMID 27870531
- [Background] Dietrich CF, Hoffmann B, Abramowicz J, Badea R, Braden B, Cantisani V, Chammas MC, Cui XW, Dong Y, Gilja OH, Hari R, Nisenbaum H, Nicholls D, Nolsoe CP, Nurnberg D, Prosch H, Radzina M, Recker F, Sachs A, Saftoiu A, Serra A, Sweet L, Vinayak S, Westerway S, Chou YH, Blaivas M. Medical Student Ultrasound Education: A WFUMB Position Paper, Part I. Ultrasound Med Biol. 2019 Feb;45(2):271-281. doi: 10.1016/j.ultrasmedbio.2018.09.017. Epub 2018 Nov 27. PMID 30497768